CLINICAL TRIAL: NCT06931951
Title: The Effectiveness and Safety of Pharmacopuncture on Inpatients With Acute Knee Pain Caused by Traffic Accidents : A Pragmatic Randomized Controlled Pilot Trial
Brief Title: The Effectiveness and Safety of Pharmacopuncture on Inpatients With Acute Knee Pain Caused by Traffic Accidents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2025-02
Record Dates: First submitted 2025-03-12; First posted 2025-04-17 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pharmacologic Action

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee Pharmacoacupuncture group (Experimental): 20 patients in the Knee Pharmacoacupuncture group
  Interventions: Procedure: Knee Pharmacoacupuncture
- Oriental medicine integrated treatment group (Active Comparator): 20 patients in the Oriental medicine integrated treatment group
  Interventions: Procedure: Oriental medicine integrated treatment

INTERVENTIONS:
Procedure: Knee Pharmacoacupuncture — Physician choose the adequate type and dose of pharmacoacupuncture and needle type
  Other Names: Drug: Herbal extract-based pharmacopuncture
  Arms: Knee Pharmacoacupuncture group
Procedure: Oriental medicine integrated treatment — Physician choose the integrated oriental medicine treatment other than herbal acupuncture.
  Other Names: Device: Acupuncture needles, cupping devices, and moxibustion devices, etc.
  Arms: Oriental medicine integrated treatment group

SUMMARY:
The purpose of this study is to reveal the effectiveness and safety of knee herbal acupuncture for patients with acute knee joint pain caused by a traffic accident. It is a practical clinical study to confirm the comparative effectiveness by comparing the strategy of treating knee herbal acupuncture in parallel with the strategy of treating it with integrated oriental medicine treatment, which is an existing treatment method.

ELIGIBILITY:
Inclusion Criteria:

* When the NRS (Numeric Rating Scale) of knee pain caused by a traffic accident is 5 or higher.
* Patients hospitalized for traffic accident treatment.
* Patients with acute pain within 14 days of experiencing knee pain due to a traffic accident.
* Patients aged between 19 and 70 years old.
* participants who agree to participate in clinical research and provide written test subject consent.

Exclusion Criteria:

* For patients diagnosed with a specific serious disease that may cause knee pain (acute fracture, dislocation, complete rupture of ligaments, etc.)
* If the cause of the pain is caused by a disease other than the knee (tumor, fibromyalgia, rheumatoid arthritis, gout, lumbar disc herniation, etc.)
* Cases where surgical intervention is required due to suspected acute fracture, dislocation, or ligament and cartilage damage
* If there is another acute disease (stroke, myocardial infarction, kidney disease, diabetic neuropathy, dementia, epilepsy, etc.) that may interfere with the treatment effect or interpretation of results
* Patients currently taking steroids, immunosuppressants, mental illness drugs, or other drugs that may affect their findings
* Inadequate or unsafe medication: hemorrhagic disease, anticoagulant therapy, severe diabetic patients with risk of infection
* Patients who have taken drugs that may affect pain, such as Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), or have received herbal acupuncture or physical therapy within the past week
* In the case of pregnant women and in the case of planning to become pregnant or nursing
* Patients within 3 months after knee surgery or if knee replacement surgery was performed
* If it has been less than 1 month since participants finished participating in another clinical study, or if participants are planning to participate in another clinical study during the study participation and follow-up period within 6 months from the date of selection
* If it is difficult to fill out the consent form for research participation
* In cases where it is difficult for other researchers to participate in clinical research

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee pain numeric rating scale (NRS) | through admission completion, an average of 1week, 2 weeks and 4 weeks after admission date
  The intensity of knee pain will be assessed using the NRS. In the NRS, participants choose a number from 0 to 10 that best describes participant's comfort (0 being no pain and 10 being the most comfortable they can imagine).

SECONDARY OUTCOMES:
Range of motion (ROM) | Enrollment date, Discharge date(On average, 1 week after admission)
  Passive ROM will be measured before and after treatment to evaluate changes before and after treatment. Passive ROM is evaluated by measuring the angle between the subject's lower extremity and an imaginary line drawn vertically from the ground at the maximum range of motion of the subject's knee joint in flexion, extension, left flexion, and right flexion. If measurement is not possible due to pain, it will be recorded as UC.
Korean Western Ontario & McMaster, K-WOMAC | Enrollment date, Discharge date(On average, 1 week after admission), 2 and 4 weeks after admission date
  K-WOMAC is a 24-item questionnaire developed to evaluate the degree of disability related to knee pain. Each question is divided into 5 levels and consists of 5 questions in the pain evaluation section, 2 questions in the stiffness evaluation section, and 17 questions in the functional disability evaluation section. The higher the score, the more severe the disability.
EuroQol-5 Dimension (EQ-5D-5L) | Enrollment date, Discharge date(On average, 1 week after admission), 2 and 4 weeks after admission date
  EQ-5D-5L is a method of evaluating health status from various aspects and then indirectly calculating the quality weight of a specific health status using pre-assigned preference scores for each functional level. It is the most widely used among several indirect measurement methods. there is. The EQ-5D-5L consists of 5 questions. Each question includes mobility, self-care, usual activities, pain/discomfort, and anxiety/depression ( Ask about the level of anxiety/depression, etc. Weights are assigned according to the level of each item, and the preference score calculation equation is presented based on these weights and constants.
Patient Global Impression of Change (PGIC) | Discharge date(On average, 1 week after admission), 2 and 4 weeks after admission date
  This is a method that allows participants to subjectively evaluate the degree of improvement on a 7-level scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Daejeon Jaseng Hospital of Korean Medicine, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No